CLINICAL TRIAL: NCT01583075
Title: Pulmonary Vein Ablation With Magnetic Navigation in Patients With Therapy-refractory Symptomatic Atrial Fibrillation: Comparison of "Single Ring" and Circumferential Ablation Techniques
Brief Title: Pulmonary Vein Ablation of Atrial Fibrillation Using Magnetic Navigation: Single Ring Versus Circumferential Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Goettingen (Other)
Collaborators: Stereotaxis (Industry)
Responsible Party: Principal Investigator, Markus Zabel, Prof. Dr. Markus Zabel, University Medical Center Goettingen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STXS 10-005
Record Dates: First submitted 2012-04-20; First posted 2012-04-23 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Pulmonary Vein Isolation, Ablation Time, Procedure Time, Freedom Form Atrial Fibrillation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Circumferential ablation (Other)
  Interventions: Procedure: Circumferential pulmonary vein ablation
- Single ring ablation (Experimental)
  Interventions: Procedure: single ring pulmonary vein ablation

INTERVENTIONS:
Procedure: Circumferential pulmonary vein ablation — Circumferential pulmonary vein ablation
  Arms: Circumferential ablation
Procedure: single ring pulmonary vein ablation — single ring pulmonary vein ablation
  Arms: Single ring ablation

SUMMARY:
The single-ring ablation method aims for isolation of the posterior LA wall including the pulmonary veins. If avoiding ablation on the posterior LA wall esophageal injury is unlikely.

Aim of this prospective study was to evaluate the safety and efficacy of an RMN-guided single-ring ablation method as compared to standard RMN-guided circumferential PVA.

ELIGIBILITY:
Inclusion Criteria:

* drug refractory AF patients undergoing PVA

Exclusion Criteria:

* drug refractory AF patients undergoing repeat PVA

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-12; Primary Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Acute procedural success | After the end of the ablation procedure
  number of PVs isolated at the end of the ablation procedure

SECONDARY OUTCOMES:
Long-term procedural success | 12 months
  long-term freedom from any AT/AF episodes

CONTACTS AND LOCATIONS:
Overall Officials: Markus Zabel, MD, Principal Investigator — Clinical Electrophysiology, University Medical Center Goettingen
Locations (1):
- UMC Göttingen, Göttingen, Lower Saxony, Germany

REFERENCES:
- [Background] Thomas SP, Lim TW, McCall R, Seow SC, Ross DL. Electrical isolation of the posterior left atrial wall and pulmonary veins for atrial fibrillation: feasibility of and rationale for a single-ring approach. Heart Rhythm. 2007 Jun;4(6):722-30. doi: 10.1016/j.hrthm.2007.01.034. Epub 2007 Feb 9. PMID 17556191